CLINICAL TRIAL: NCT02186392
Title: The Impact of Ergonomic Circadian Light on Hospitalized Stroke Patients in a Rehabilitation Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Helle Klingenberg Iversen, MD, DmSc, MD, DMSc, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-4-2013-114
Record Dates: First submitted 2014-06-03; First posted 2014-07-10 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Stroke; Sleep Apnea Syndromes; Depression; Anxiety
Keywords: Depression; Anxiety; Stroke; Cerebral Infarction; Sleep disorders; Circadian Rhythm disorders; Circadian Light; Light therapy; Melatonin; Sleep; Sleep apnea; Coagulation disturbances; Bone metabolism; Rehabilitation; Mood disorders; Mental disorders; Neurologic Manifestations; Signs and Symptoms Cerebrovascular Disorders; Brain Diseases; Vascular Disease; Brain Infarction; Brain Ischemia
MeSH Terms: conditions — Stroke; Sleep Apnea Syndromes; Depression; Anxiety Disorders; Cerebral Infarction; Sleep Wake Disorders; Chronobiology Disorders; Mood Disorders; Mental Disorders; Neurologic Manifestations; Brain Diseases; Vascular Diseases; Brain Infarction; Brain Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control department (No Intervention): The control department where the conventional light is installed.
- Circadian Light luminaries (Experimental): The department where the special circadian light is installed. The light is programmed to have the desired light intensity (lux), color temperature (Kelvin) and wavelength (nm) according to the knowledge about the phase-response curve.
  Interventions: Device: Circadian Light luminaries

INTERVENTIONS:
Device: Circadian Light luminaries — The light is programmed to have the desired light intensity (lux), color temperature (Kelvin) and wavelength (nm) according to the knowledge about the phase-response curve.
  Other Names: Chroma Viso; Ergonomic
  Arms: Circadian Light luminaries

SUMMARY:
The purpose of this study is to investigate the impact of exposure to ergonomic circadian light on physiological and mental parameters in stroke patients admitted for rehabilitation.

DETAILED DESCRIPTION:
Stroke annually affects approximately 12,000 Danes and there are approximately 50,000 living persons with sequelae after stroke in Denmark. Stroke is the major cause of acquired cerebral disability among adults and the second most common cause of dementia and the third leading cause of death.

Besides the acute stroke treatment, an effective rehabilitation program is necessary for optimal recovery. A prerequisite for this is that stroke patients are able to contribute optimally to the training, however, changes in the sleep pattern and disturbed circadian rhythm may exert negative effects.

Little is known about circadian disturbances in relation to rehabilitations and which consequences it may have on the physiological and mental levels.

The investigators will investigate the following hypotheses:

A: Ergonomic circadian light improves well-being and fatigue in post-stroke patients compared with a control group receiving standard light facilities.

B: Ergonomic circadian light induces improve sleep-wake cycle and circadian rhythm in post-stroke patients compared with a control group receiving standard light facilities.

C: Ergonomic circadian light induces reduction in depression and anxiety in post-stroke patients compared with a control group receiving standard light facilities.

D: Ergonomic circadian light improves the cognitive function in post-stroke patients compared with a control group receiving standard light facilities.

E: Ergonomic circadian light induces reduction in autonomic dysfunction in post-stroke patients compared with a control group receiving standard light facilities.

F: Ergonomic circadian light will regulate circadian rhythm specific blood tests in post-stroke patients compared with a control group receiving standard light facilities.

From the acute stroke unit the patients will be random transferred to two rehabilitation units where the will be the intervention unit with the circadian light installed and a control unit with conventional light.

At the inclusion, patients will be assessed by the following interventions mentioned below, which again will be evaluated at discharge. The incompetent patients to these interventions must abstain.

The numbers of patients who are expected to be included are 110 calculated with 25% dropout resulting in approximately 80 patients.

All patients who are found suitable for admission to the two rehabilitation departments will be listed. If a patient is not suitable for inclusion in the study the reason will be described and published.

During hospitalization on the rehabilitation unit following tests/interventions will be performed on the patients:

* Stroke classification
* Sleep physiology
* Sleep biochemistry
* Test for depression
* Test for cognitive function
* Test for anxiety
* Test Fatigue
* Testing for sleep quality
* Test for Quality of well being
* Chronotype classification
* Autonomic dysfunction
* Status of physical rehabilitation
* Functional MRI Resting state
* Circadian blood samples
* Ophthalmological examination

ELIGIBILITY:
Inclusion Criteria:

* Patients evaluated as candidates to the rehabilitation units from May 1th 2014 to May 1th 2015.

Exclusion Criteria:

* Glasgow Coma Scale (GCS) < 15
* No functioning of the optic nerve or retina in both eyes
* Unable to open both eyes
* Non communicating patients e.g. aphasia (incompetent patients)
* Unable to cooperate to the physical examinations
* Less than 2 weeks of hospitalization in the rehabilitation department
* If the sub investigator finds the study participant unfit to conduct the investigations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
well-being | The participants will be tested at the inklusion (1-2 days before admission to the rehabilitation unit) and at discharge. A hospital stay with an average duration of about 4 weeks.
  The test will be performed at the admission for the rehabilitation unit and at discharged.
  Well-being and fatigue is according to WHO-5 well-being scale, Multidimensional Fatigue Inventory-20 (MFI-20), Visual Analog Scala for fatigue.
Depression | The participants will be tested at the inklusion (1-2 days before admission to the rehabilitation unit) and at discharge. A hospital stay with an average duration of about 4 weeks.
  The test will be performed at the admission for the rehabilitation unit and at discharged.
  Mild, moderate or severe depression according to Hamilton-D6 (HAM-D6), Major Depression Inventory (MDI) or Hospital Anxiety and Depression Scale (HADS).
Anxiety | The participants will be tested at the inklusion (1-2 days before admission to the rehabilitation unit) and at discharge. A hospital stay with an average duration of about 4 weeks.
  The test will be performed at the admission for the rehabilitation unit and at discharged.
  Anxiety according to HADS.
Circadian rhythm specific blood marker | The participants will be tested at the inklusion (1-2 days before admission to the rehabilitation unit) and at discharge. A hospital stay with an average duration of about 4 weeks.
Sleep and sleep-wake cycle | The participants will be tested at the inklusion (1-2 days before admission to the rehabilitation unit) and at discharge. A hospital stay with an average duration of about 4 weeks.
  The test will be performed at the admission for the rehabilitation unit and at discharged.
  Sleep will be measured according to Polysomnography, Actigraph, Pittsburgh Sleep Quality Index (PSQI) and Epworth Sleepiness Scale.

SECONDARY OUTCOMES:
Cognitive function | The participants will be tested at the inklusion (1-2 days before admission to the rehabilitation unit) and at discharge. A hospital stay with an average duration of about 4 weeks.
  The test will be performed at the admission for the rehabilitation unit and at discharged.
  Level of cognitive function is according to Montreal Cognitive Assessment (MoCA), Trail Marking Test (TMT), and Confusion Assessment Method.
Autonomic function | The participants will be tested at the inklusion (1-2 days before admission to the rehabilitation unit) and at discharge. A hospital stay with an average duration of about 4 weeks.
  The test will be performed at the admission for the rehabilitation unit and at discharged.
  autonomic dysfunction will be measured according to Polysomnography by heart rate and blod pressure.

OTHER OUTCOMES:
Physical status | The participants will be tested at the inklusion (1-2 days before admission to the rehabilitation unit) and at discharge. A hospital stay with an average duration of about 4 weeks.
  The test will be performed at the admission for the rehabilitation unit and at discharged.
  Physical status/testing for mobilization will be according to Barthel Index, Motor Assessment Scale, 10-meters walk test, National Institutes of Health Stroke Scale (NIHSS) and Modified Rankin Scale (mRS).
Stroke classification | The participants will be tested at the inklusion (1-2 days before admission to the rehabilitation unit) and at discharge. A hospital stay with an average duration of about 4 weeks.
  Stroke classification according to TOAST criteria and Oxfordshire criteria.
Ophthalmological status | during hospitalization in the rehabilitation unit.
  Ophthalmological status will be measured according to optical coherence tomography, fundus photography, pupillometry, visual acuity, color vision, intraocular pressure, Slitlamp examination and grading of the lens.
cause of death after stroke | assessed at follow-up during admission

CONTACTS AND LOCATIONS:
Overall Officials: Helle K Iversen, MD, DMSc, Study Chair — Department of clinical stroke reseach, Department of Neurology, Glostrup Hospital.; Poul Jennum, MD, DMSc, Study Director — Department Director of Danish Center for Sleep Medicine, Neurophysiological Department, Glostrup Hospital.; Anders S West, MD, Principal Investigator — Department of clinical stroke reseach, Department of Neurology, Glostrup Hospital.
Locations (1):
- Department of clinical stroke reseach, Department of Neurology, Glostrup Hospital., Glostrup Municipality, Denmark